CLINICAL TRIAL: NCT00576706
Title: A Phase III, Randomized, Double-dummy, Double Blind, Misoprostol-comparative Clinical Trial to Evaluate the Efficacy and Safety of Mucosta® Tablet in the Prevention of NSAID-induced Gastrointestinal Complications
Brief Title: PReventive Efficacy and Safety of rEbamipide on Nsaid Induced Mucosal Toxicity
Acronym: PRESENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Korea Otsuka Pharmaceutical Co.,Ltd., Korea Otsuka Pharmaceutical Co.,Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 037-KOA-0701i
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Ankylosing Spondylitis
Keywords: Patients with rheumatoid arthritis, osteoarthritis, and ankylosing spondylitis or any other arthritis-like disease requiring continuous NSAIDs therapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Spondylitis, Ankylosing | interventions — rebamipide; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rebamipide
- 2 (Active Comparator)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Rebamipide — Rebamipide 100㎎, 12 weeks
  Other Names: Mucosta
  Arms: 1
Drug: Misoprostol — Misoprostol 200㎍ 12 weeks
  Other Names: Cytotec®
  Arms: 2

SUMMARY:
To prove that the efficacy and safety of Mucosta® (Rebamipide) is non-inferior to those of Cytotec® (Misoprostol), in terms of prevention of NSAID-induced gastric ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent after being informed of the clinical trial
2. Males or females 19 years of age
3. Intake of any brand of NSAIDs in more than half of daily dose for at least the previous 4 weeks.

Exclusion Criteria:

1. Necessary to proceed in concomitant treatment with epileptic medications, anti-chollinergics, prokinetics, sucralfate
2. Presence or history of allergic drug reaction to the following medications; rebamipide, Misoprostol, NSAIDs designated to the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of gastric ulcer on gastroendoscopy result at 12-week | 12 weeks

SECONDARY OUTCOMES:
Rate of Therapeutic failure | 12 weeks
Severity of gastrointestinal symptoms | 12 weeks
Antacid consumption | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Heon Park, MD PhD, Principal Investigator — Catholic University Hospital
Locations (10):
- South Korea (10):
  - Bucheon-si
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Jeonju
  - Jinju
  - Pusan
  - Seoul
  - Suwon